CLINICAL TRIAL: NCT04260724
Title: Prospective, Randomized, Evaluator-blind, Single Center Study on the Effect of Transcranial Magnetic Stimulation in Mild to Moderate Alzheimer's Disease
Brief Title: Study on the Effect of Transcranial Magnetic Stimulation in Mild to Moderate Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Duk Lyul Na, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMC_2019-04-010-004
Record Dates: First submitted 2020-01-22; First posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Mild to Moderate Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMS group (Active Comparator): Transcranial magnetic stimulation for four weeks
  Interventions: Device: TMS
- Sham group (Sham Comparator): sham coil stimulation for four weeks (Although the sound of sham coil is the same to that of real TMS during intervension, no stimulation is applied. )
  Interventions: Device: sham coil stimulation

INTERVENTIONS:
Device: TMS — * stimulation intensity : motor threshold 100%
  * stimulation frequency : 1600 pulses for 20 minutes
  * stimulation duration :for four weaks, 20 minutes/day, 5 days per week (Monday - Friday )
  Arms: TMS group
Device: sham coil stimulation — no stimulation Although the sound from device during stimulation is similar, no stimulation is applied.
  Arms: Sham group

SUMMARY:
The investigators will compare cognitition, mood (depression), ADL, and brain structural and functional MRI before and after 4-week transcranial magnetic stimulation in patients with mild to moderate Alzheimer's disease.

The investigators also compare the change of cognitition, mood (depression), ADL, and brain structural and functional MRI between TMS group and sham coil group.

DETAILED DESCRIPTION:
Each 16 patients will be allocated to TMS group and sham coil group. Before TMS/sham coil stimulation, the investigators will take fMRI of each patient, and figure out which focus has strongest connectivity to hippocampus among lateral parietal regions of the brain. The investigators will fix the TSM transduced and apply accurate TMS stimulation to the focus using personalized frames. The investigators will make the frame using 3D printing technology.

After 4 week- TMS stimulation, the investigators will compare cognitition, mood (depression), ADL, and brain structural and functional MRI beween baseline and after intervention. The investigators also compare the change of cognitition, mood (depression), ADL, and brain structural and functional MRI between TMS group and sham coil group.

ELIGIBILITY:
Inclusion Criteria:

* patients who visited memory clinic of Samsung Medical Center
* aged 55 ~ 90
* diagnosed as probable Alzheimer dementia according to NIA-AA guideline 2011, or MCI patiens with amyloid PET positivity
* below -1SD in SVLTdelayed recall test and RCFT delayed recall test
* K-MMSE >=18
* no epileptic discharge in EEG
* no history of epilepsy
* no arrhythmia or MI in ECG
* can read and write Korean (literate)
* volunteer and agree to the registration

Exclusion Criteria:

* no other neurologic deficit which can cause dementia except for Alzheimer's disease
* paitient who has severe cerebral white matter hyperintensities. (deep white matter >=2.5cm and caps or band >=1.0 cm)
* patients with severe medical disease including caner and ishemic heart disease
* claustrophobia or allergic to contrast of MRI
* medical deviced which is not removable (e.g pacemaker, cochlear implantation, dental prosthesis)
* history of brain surgery, and intervension or surgery of intra/extracranial artery(e.g. carotid artery stent insertion, CEA)
* patient with dyspnea during resting
* history of loss of consciousness for more than 1 hour except for general anesthesia
* patients who cannot read written material because of poor visual acuity
* patients who cannot communicate because of severe hearing difficulty
* history of ototoxicity medication or exposure severe noises
* determined as inapropriate to participate clinical trial

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-02-07 (Estimated); Primary Completion 2021-02-07 (Estimated); Study Completion 2022-02-07 (Estimated)

PRIMARY OUTCOMES:
the short term change of K-MMSE score in TMS group | 4 weeks
  the short term change of K-MMSE (Korean version of mini mental status exam) score in TMS group
the short term change of K-MoCA score in TMS group | 4 weeks
  the short term change of K-MoCA (Korean version of Montreal cognitive assessment) score in TMS group
the short term change of ADAS-Cog score in TMS group | 4 weeks
  the short term change of ADAS-Cog(the Alzheimer's disease assessment scale-cognitive subscale) score in TMS group
the short term change of COWAT score in TMS group | 4 weeks
  the short term change of COWAT(controlled oral word association) score in TMS group
the short term change of Stroop score in TMS group | 4 weeks
  the short term change of Stroop score in TMS group
the short term change of TMT score in TMS group | 4 weeks
  the short term change of TMT(trail-making test) score in TMS group
the short term change of RVP score in TMS group | 4 weeks
  the short term change of RVP(raid visual information processing) score in TMS group
the short term change of SWM score in TMS group | 4 weeks
  the short term change of SWM (spatial working memory) score in TMS group
the short term change of PRM score in TMS group | 4 weeks
  the short term change of PRM(pattern recognition memory) score in TMS group

SECONDARY OUTCOMES:
the long term change of K-MMSE score in TMS group | 8 weeks
  the long term change of K-MMSE (Korean version of mini mental status exam) score in TMS group
the long term change of K-MoCA score in TMS group | 8 weeks
  the long term change of K-MoCA (Korean version of Montreal cognitive assessment) score in TMS group
the long term change of ADAS-Cog score in TMS group | 8 weeks
  the long term change of ADAS-Cog(the Alzheimer's disease assessment scale-cognitive subscale) score in TMS group
the long term change of COWAT score in TMS group | 8 weeks
  the long term change of COWAT(controlled oral word association) score in TMS group
the long term change of Stroop score in TMS group | 8 weeks
  the long term change of Stroop score in TMS group
the long term change of TMT score in TMS group | 8 weeks
  the long term change of TMT(trail-making test) score in TMS group
the long term change of RVP score in TMS group | 8 weeks
  the long term change of RVP(raid visual information processing) score in TMS group
the long term change of SWM score in TMS group | 8 weeks
  the long term change of SWM (spatial working memory) score in TMS group
the long term change of PRM score in TMS | 8 weeks
  the long term change of PRM(pattern recognition memory) score in TMS group
the change of ADL(activity of daily life) in TMS group | 4 weeks
  the score change of S-IADL(Seoul-Instrumental activities of daily life)
the short term change of mood (depression) in TMS group | 4 weeks
  the score change of GDS(geriatric depression scale) short form
the long term change of mood (depression) in TMS group | 8 weeks
  the score change of GDS(geriatric depression scale) short form
the change of brain function in TMS group | 4 weeks
  the qualititve change of resting functional MRI
the change of brain structure in TMS group | 4 weeks
  the change of FA (fractional anisotropy) value in DTI (diffusion tensor imaging) analysis
the comparison of short term change of K-MMSE score between TMS group and sham group | 4 weeks
  the score change of K-MMSE (Korean version of mini mental status exam)
the comparison of short term change of K-MoCA score between TMS group and sham group | 4 weeks
  the score change of K-MoCA (Korean version of Montreal cognitive assessment)
the comparison of short term change of CDR-SOB between TMS group and sham group | 4 weeks
  the score change of CDR-SOB (Clinical dementia rating-sum of boxes)
the comparison of short term change of ADAS-Cog between TMS group and sham group | 4 weeks
  the score change of ADAS-Cog ( the Alzheimer's disease assessment scale-cognitive subscale)
the comparison of short term change of COWAT score between TMS group and sham group | 4 weeks
  the score change of COWAT(controlled oral word association) score
the comparison of short term change of Stroop test score between TMS group and sham group | 4 weeks
  the score change of Stroop test score
the comparison of short term change of TMT between TMS group and sham group | 4 weeks
  the score change of TMT (trail making test)
the comparison of short term change of RVP score between TMS group and sham group | 4 weeks
  the score change of RVP(raid visual information processing) score
the comparison of short term change of SWM between TMS group and sham group | 4 weeks
  the score change of SWM (spatial working memory) score
the comparison of short term change of PRM between TMS group and sham group | 4 weeks
  the score change of PRM(pattern recognition memory) score
the comparison of change of K-MMSE between TMS group and sham group | 8 weeks
  the score change of K-MMSE(Korean version of mini mental status exam)
the comparison of long term change of K-MoCA between TMS group and sham group | 8 weeks
  the score change of K-MoCA (Korean version of Montreal cognitive assessment)
the comparison of long term change of CDR-SOB between TMS group and sham group | 8 weeks
  the score change of CDR-SOB(Clinical dementia rating-sum of boxes)
the comparison of long term change of ADAS-Cog between TMS group and sham group | 8 weeks
  the score change of ADAS-Cog ( the Alzheimer's disease assessment scale-cognitive subscale)
the comparison of long term change of COWAT score between TMS group and sham group | 8 weeks
  the score change of COWAT(controlled oral word association) score
the comparison of long term change of stroop test score between TMS group and sham group | 8 weeks
  the score change of stroop test score
the comparison of long term change of TMT score between TMS group and sham group | 8 weeks
  the score change of TMT(trail making test)
the comparison of long term change of RVP score between TMS group and sham group | 8 weeks
  the score change of RVP(raid visual information processing)
the comparison of long term change of SWM score between TMS group and sham group | 8 weeks
  the score change of SWM (spatial working memory) score
the comparison of long term change of cognitive function between TMS group and sham group | 8 weeks
  the score change of PRM(pattern recognition memory) score
the comparison of short term change of mood (depression) between TMS group and sham group | 4 weeks
  the score change of GDS (geriatric depression scale) short form
the comparison of long term change of mood (depression) between TMS group and sham group | 8 weeks
  the score change of GDS (geriatric depression scale) short form
the comparison of short term change of ADL between TMS group and sham group | 4 weeks
  the score change of S-IADL(Seoul instrumental activity of daily life )
the comparison of long term change of ADL between TMS group and sham group | 8 weeks
  the score change of S-IADL(Seoul instrumental activity of daily life )
the comparison of change of resting fMRI between TMS group and sham group | 4 weeks
  the qualititve change of resting fMRI
the comparison of change of FA value between TMS group and sham group | 4 weeks
  the change of FA(fractional anisotropy) value in DTI(diffusion tensor imaging) analysis

CONTACTS AND LOCATIONS:
Overall Officials: Duk L Na, MD PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nilakantan AS, Mesulam MM, Weintraub S, Karp EL, VanHaerents S, Voss JL. Network-targeted stimulation engages neurobehavioral hallmarks of age-related memory decline. Neurology. 2019 May 14;92(20):e2349-e2354. doi: 10.1212/WNL.0000000000007502. Epub 2019 Apr 17. PMID 30996057
- [Background] Cotelli M, Manenti R, Cappa SF, Geroldi C, Zanetti O, Rossini PM, Miniussi C. Effect of transcranial magnetic stimulation on action naming in patients with Alzheimer disease. Arch Neurol. 2006 Nov;63(11):1602-4. doi: 10.1001/archneur.63.11.1602. PMID 17101829
- [Background] Cotelli M, Calabria M, Manenti R, Rosini S, Zanetti O, Cappa SF, Miniussi C. Improved language performance in Alzheimer disease following brain stimulation. J Neurol Neurosurg Psychiatry. 2011 Jul;82(7):794-7. doi: 10.1136/jnnp.2009.197848. Epub 2010 Jun 23. PMID 20574108
- [Background] Cotelli M, Manenti R, Cappa SF, Zanetti O, Miniussi C. Transcranial magnetic stimulation improves naming in Alzheimer disease patients at different stages of cognitive decline. Eur J Neurol. 2008 Dec;15(12):1286-92. doi: 10.1111/j.1468-1331.2008.02202.x. PMID 19049544
- [Background] Wang JX, Rogers LM, Gross EZ, Ryals AJ, Dokucu ME, Brandstatt KL, Hermiller MS, Voss JL. Targeted enhancement of cortical-hippocampal brain networks and associative memory. Science. 2014 Aug 29;345(6200):1054-7. doi: 10.1126/science.1252900. PMID 25170153
- [Background] Koch G, Bonni S, Pellicciari MC, Casula EP, Mancini M, Esposito R, Ponzo V, Picazio S, Di Lorenzo F, Serra L, Motta C, Maiella M, Marra C, Cercignani M, Martorana A, Caltagirone C, Bozzali M. Transcranial magnetic stimulation of the precuneus enhances memory and neural activity in prodromal Alzheimer's disease. Neuroimage. 2018 Apr 1;169:302-311. doi: 10.1016/j.neuroimage.2017.12.048. Epub 2017 Dec 19. PMID 29277405
- [Background] Ridding MC, Rothwell JC. Is there a future for therapeutic use of transcranial magnetic stimulation? Nat Rev Neurosci. 2007 Jul;8(7):559-67. doi: 10.1038/nrn2169. PMID 17565358
- [Background] Bondi MW, Edmonds EC, Jak AJ, Clark LR, Delano-Wood L, McDonald CR, Nation DA, Libon DJ, Au R, Galasko D, Salmon DP. Neuropsychological criteria for mild cognitive impairment improves diagnostic precision, biomarker associations, and progression rates. J Alzheimers Dis. 2014;42(1):275-89. doi: 10.3233/JAD-140276. PMID 24844687
- [Background] Weissman MM, Myers JK, Tischler GL, Holzer CE 3rd, Leaf PJ, Orvaschel H, Brody JA. Psychiatric disorders (DSM-III) and cognitive impairment among the elderly in a U.S. urban community. Acta Psychiatr Scand. 1985 Apr;71(4):366-79. doi: 10.1111/j.1600-0447.1985.tb02536.x. PMID 4003102
- [Result] Kim S, Nilakantan AS, Hermiller MS, Palumbo RT, VanHaerents S, Voss JL. Selective and coherent activity increases due to stimulation indicate functional distinctions between episodic memory networks. Sci Adv. 2018 Aug 22;4(8):eaar2768. doi: 10.1126/sciadv.aar2768. eCollection 2018 Aug. PMID 30140737
- [Derived] Jung YH, Jang H, Park S, Kim HJ, Seo SW, Kim GB, Shon YM, Kim S, Na DL. Effectiveness of Personalized Hippocampal Network-Targeted Stimulation in Alzheimer Disease: A Randomized Clinical Trial. JAMA Netw Open. 2024 May 1;7(5):e249220. doi: 10.1001/jamanetworkopen.2024.9220. PMID 38709534